CLINICAL TRIAL: NCT06705907
Title: Improving Academic and Social Functioning in Middle-Schoolers With Autism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB#2024-0148; 1R01HD113534-01A1 (NIH)
Record Dates: First submitted 2024-11-23; First posted 2024-11-26 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: social skills; executive functions; academic achievement; middle school
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Social Skills | interventions — Schools

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Achieving Independence & Mastery in School (AIMS) (Experimental): AIMS targets executive functioning skills using evidence-based strategies for youth with ASD to promote increased independence related to academics. Each session involves a review of a real world practice assignment and a didactic component illustrating key concepts followed by an in-session practice of the key concepts and strategies with coaching from a therapist. A behavior agreement is used to identify specific goals for adolescents to work on in collaboration with their caregivers and specific rewards earned for meeting their goals. Adolescents are assigned a real world practice assignment each session that consists of additional practice of strategies to further build and generalize skills between sessions.
  Interventions: Behavioral: Achieving Independence and Mastery in School (AIMS)
- Building Essential Social Skills for Teens (BESST) (Active Comparator): BESST targets social skills using evidence-based strategies and includes sessions related to starting, joining, maintaining, and ending conversations and making, maintaining, and deepening friendships. Each skill will be introduced in a didactic lesson which includes modeling of the targeted skill by a therapist. Adolescents will role-play new skills during the session before receiving a homework assignment to practice the skill at home. Caregivers will receive training in social-communication difficulties in ASD and suggestions for supporting development of these skills. The sessions are specifically focused on generalizing newly learned skills to both home and school.
  Interventions: Behavioral: Building Essential Social Skills for Teens (BESST)

INTERVENTIONS:
Behavioral: Achieving Independence and Mastery in School (AIMS) — Intervention targeting academic executive functioning
  Other Names: AIMS
  Arms: Achieving Independence & Mastery in School (AIMS)
Behavioral: Building Essential Social Skills for Teens (BESST) — Intervention targeting social skills
  Other Names: BESST
  Arms: Building Essential Social Skills for Teens (BESST)

SUMMARY:
The goal of this study is to test how well two group interventions work for middle-school children with Autism Spectrum Disorder (ASD). One of the interventions focuses on teaching parents and adolescent skills to help improve their social functioning and the other focuses on teaching parents and adolescents skills to improve organization, planning, and study skills. Eligible participants will be randomly (like a coin flip) assigned to attend one of the two interventions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism
* No intellectual disability
* Problems with organization, materials management, and planning and prioritization
* Problems with social skills
* Fully included in middle school
* Stable medication and behavioral treatment regime

Exclusion Criteria:

* Home schooled
* Severe co-occurring psychopathology (e.g., aggression, suicidal)
* Non English-speaking

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 224 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Behavior Rating Inventory of Executive Functioning, 2nd Edition | From enrollment to the end of treatment at 8 weeks.
  The BRIEF-2 assesses real-world EF behaviors in the home and school environments.
  The T-scores range from 30:99 with higher scores being worse.
Homework Problems Checklist | From enrollment to end of treatment at 8 weeks.
  The HPC assesses Homework Completion and Homework Management. Scores for Homework Completion range from 0 to 36 and for Homework Management from 0 to 21. Lower scores are better.
Academic Performance Rating Scale | From enrollment to end of treatment at 8 weeks.
  The teacher-completed APRS assesses how well the adolescent is performing academically with 3 subscales (Academic Success, Academic Productivity, and Impulse Control). The two scores to be used in the current study include the Academic Success score which ranges from 7 to 35, while the Academic Productivity score ranges from 12 to 60. Higher scores are better.

SECONDARY OUTCOMES:
Children's Organizational Skills Scale | From enrollment to the end of treatment at 8 weeks.
  The COSS is a psychometrically strong rating scale assessing Organized Actions, Task Planning, and Memory & Materials Management. The T scores for each subscale range from 20 to 83 and higher scores indicate worse functioning.
Weekly Calendar Planning Activity | From enrollment to the end of treatment at 8 weeks.
  The WCPA is an objective measure of metacognition (i.e., planning, inhibition, problem solving, keeping track of rules, and monitoring passage of time) while performing a multiple-step activity (i.e., scheduling multiple appointments while adhering to various rules). The WCPA will report total appointments entered (0 to 10) and total correct appointments entered (0 to 10) with higher values being better.
Social Skills Assessment (TRIAD) | From enrollment to the end of treatment at 8 weeks.
  The TRIAD assesses social skills (i.e., emotion understanding and perspective taking, initiating and ending interactions, responding to others, maintaining interactions and problem solving, and following social rules) rated on a 1 to 4 scale (1=not very well to 4=very well). Items rated 2 or less are considered areas of weakness. Items rated as 3 or above are considered areas of strength.

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Tamm, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati; Amie Duncan, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be entered into NIMH's Data Archive (NDA) in order to contribute to the advancement of research on individuals with ASD. In our Background History Form, we will collect the prerequisite information (i.e., specific information such as legal name, date of birth, sex, and city of birth) needed to generate a GUID. Informed consent documents will inform participants that their data will be entered into NDA.
Supporting Information: Study Protocol, ICF
Time Frame: August 31, 2029
Access Criteria: Investigators interested in using the data obtained in this study will be directed to obtain the data from NDA. Other materials can be obtained from the study principal investigators upon reasonable request.